CLINICAL TRIAL: NCT03822221
Title: What is the Best Joint Angle of the Knee and Hip to Optimize the Neuromuscular and Tendinous Adaptations Induced by Neuromuscular Electrical Stimulation of the Femoral Quadriceps? Implications for Rehabilitation
Brief Title: Angles of Knee and Hip Joints for Optimization of Neuromuscular Electrical Stimulation of the Quadriceps Femoris Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Brasilia (Other)
Collaborators: University of Burgundy (Other)
Responsible Party: Principal Investigator, João Luiz Q. Durigan, Physical Therapist, Assistant Professor, University of Brasilia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: CAAE: 94388718.8.0000.8093
Record Dates: First submitted 2018-12-07; First posted 2019-01-30 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Electrical Stimulation
Keywords: Quadriceps muscle; Electrical Stimulation; Patellar Tendon; Ultrasonography; Electromyography

STUDY DESIGN:
Intervention Model Description: After a familiarization session, there will be four sessions for testing the electrical stimulation at four different combinations of hip and knee angles for isometric contractions. The order of the combinations will be randomized, and a washout period of seven days will be reacquired between each session.
Who Masked: Participant, Outcomes Assessor
Masking Description: Volunteers will be blinded to the study hypothesis and the reason for positioning changes during the study. One researcher will be blinded for outcomes statistics analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- SK20º (Experimental): MVIC and NMES with hip at 85º and knee at 20º
  Interventions: Other: MVIC and NMES with hip at 85º and knee at 20º
- SK60º (Experimental): MVIC and NMES with hip at 85º and knee at 60º
  Interventions: Other: MVIC and NMES with hip at 85º and knee at 60º
- LK20º (Experimental): MVIC and NMES with hip at 0º and knee at 20º
  Interventions: Other: MVIC and NMES with hip at 0º and knee at 20º
- LK60º (Experimental): MVIC and NMES with hip at 0º and knee at 60º
  Interventions: Other: MVIC and NMES with hip at 0º and knee at 60º

INTERVENTIONS:
Other: MVIC and NMES with hip at 85º and knee at 20º — With hip joint at 85º (seated) and knee at 20º (SK20º), subjects will be submitted to maximal isometric voluntary contractions (15-18 per session) and to contractions evoked by neuromuscular electrical stimulation (15-18 per session).
  Arms: SK20º
Other: MVIC and NMES with hip at 85º and knee at 60º — With hip joint at 85º (seated) and knee at 60º (SK60º), subjects will be submitted to maximal isometric voluntary contractions (15-18 per session) and to contractions evoked by neuromuscular electrical stimulation (15-18 per session).
  Arms: SK60º
Other: MVIC and NMES with hip at 0º and knee at 20º — With hip joint at 0º (lying) and knee at 20º (LK20º), subjects will be submitted to maximal isometric voluntary contractions (15-18 per session) and to contractions evoked by neuromuscular electrical stimulation (15-18 per session).
  Arms: LK20º
Other: MVIC and NMES with hip at 0º and knee at 60º — With hip joint at 0º (lying down) and knee at 60º (LK60º), subjects will be submitted to maximal isometric voluntary contractions (15-18 per session) and to contractions evoked by neuromuscular electrical stimulation (15-18 per session).
  Arms: LK60º

SUMMARY:
Introduction: The muscle contractile effectiveness is influenced by the neural activation of the motor units, as well as its architecture and the elasticity of the myotendinous junction. In addition, tendinous properties also affect the production of muscle strength and function. Neuromuscular electrical stimulation (NMES) is a wide-used tool in rehabilitation for motor relearning, to reduce muscular atrophy, pain control and to improve functional performance. Although studies have demonstrated the efficacy of NMES in various clinical situations, the best joint angle (ideal muscle length) to enhance neuromuscular and tendinous adaptations induced by NMES has to be determined.

Objective: To investigate the effect of NMES on different hip and knee angles on knee extensor torque, quadriceps muscle electromyographic activity, architecture, and tendon-aponeurosis complex elongation, and tendinous properties of the patellar tendon.

Material and Methods: This is a crossover study with healthy males, aged 18-35 years. The independent variables will be: 1) NMES in different lower limb positions: knee joint angulation at 20º or 60º with hip at 0º or 80º (four combinations). The dependent variables will be: knee extensor torque, surface muscle electrical activity, muscle architecture (muscle thickness, pennation angle and fascicular length), the elongation of the tendon-aponeurosis complex of the quadriceps muscle components, and the properties (stiffness, Young's modulus and cross-sectional area) of the patellar tendon. The descriptive and analytical statistics will be carried out with measures of central tendency and dispersion, inference tests, tables and graphs. The normality of the data will be verified with the Shapiro-Wilk test. For the data that present normal distribution, the Two-Way ANOVA will be applied to verify differences among the measurements, with post-hoc of Bonferroni. The non-parametric option will be the Friedman test. Correlation coefficients will be calculated using the Pearson (parametric) or Spearman (non-parametric) correlation test. The level of statistical significance will be p <0.05.

Expected results: The effect of an NMES session on the neural, muscular and tendon adaptations related to the angular specificity of the hip and knee, indicating greater potential for strength and muscle mass gains, will be shown, which is fundamental in the prescription of electrostimulation in rehabilitation.

DETAILED DESCRIPTION:
Neuromuscular electrical stimulation (NMES) is used in various contexts due to its benefits related to motor learning, preservation of denervated muscles, training in non-cooperative / sedated individuals, pain control and relief, and improvement of athletes, young, and elderly functional performance, besides people with severe cardiopulmonary disease. Even with the solid accumulated knowledge about NMES, its potential is not fully understood, with questions to be clarified for the achievement of greater effectiveness by clinicians and scientists in the various possibilities of application.

The effects of NMES have not been determined yet in quadriceps femoris muscle in different lengths, which can be accomplished by changing the angle of the joint or joints it crosses (hip and knee). There is probably only one trial (Fahey et al., 1984) addressing this issue. In the study, two positions were compared: knee and hip extended versus knee (65º) and hip (angle not mentioned) flexed, although the purpose of the study was to evaluate only the influence of knee position. Authors found that NMES can increase isometric and isokinetic strength, but that it may be more effective to improve isokinetic performance if knee is flexed during treatment. Questions are then raised because groups were tested only with knee flexed and not also extended, and because the change in hip angle probably influenced the results. This study was also the only one found by Bax et al. (2005).

Justificative: NMES is an established tool applied as the main or an supplementary treatment in rehabilitation programs. It is necessary to establish the influence of lower limb position in the outcomes. Therefore, this study will address for the first time the effects of NMES on quadriceps voluntary and evoked strength, electrical activity, architecture, and tendon properties.

Hypothesis: In healthy young adults, the variation of the hip and knee joint angle for NMES may affect the knee extensor torque, quadriceps muscle electromyographic activity, architecture, and tendon-aponeurosis complex elongation, and tendinous properties of the patellar tendon. These factors will be facilitated when the participants are seated with the knee at 60º flexion. On the other hand, when the quadriceps is more elongated (lying with knee at 60º) or shortened (dorsal decubitus or sitting with knee extended (0º), such adaptations will not be significant.

Methods: This is a crossover trial with healthy young male subjects. The procedures will be performed in the Neuromuscular Performance Laboratory of the Faculty of Ceilândia / University of Brasília and in the Force Laboratory of the Faculty of Physical Education / University of Brasília. Subjects will perform 5 visits to the laboratory (the first visit will be a familiarization session to test NMES in each position), with a minimum interval of 48 hours between visits. Volunteers will be informed of all the procedures, purposes, benefits, and risks of the study and will sign an informed consent form before participation (the project was approved by the University Research Ethics Committee N 99221818.9.0000.0029)

* Maximal Voluntary Isometric Contraction (MVIC): An isokinetic dynamometer will be used for recording torque. The equipment axis will be visually aligned with the axis of the knee (lateral epicondyle of the femur). The lever arm of the force transducer will be firmly attached 2-3 cm above the lateral malleolus with a strap. Angulations of hip and knee will be adjusted with a goniometer. Subjects will be firmly stabilized to the chair with belts across the chest and pelvic girdle to minimize body movement. Individuals will be instructed to cross their arms with hands on shoulders and extend the knee against the strap "by pushing gradually for 3 s (ramping contraction) up to the maximum force, maintaining it for 4 s, and then decrease de amount of force gradually for more 3 s". The number of contractions will correspond to the number of ultrasound evaluations: 4 muscles (rectus femoris and the three vastus) + proximal patellar tendon + distal patellar tendon x 3 measurements for each = 18, each one separated by 1 min of rest.
* Neuromuscular electrical stimulation (NMES): NMES will be used to produce a maximal electrically evoked isometric torque, which will be assessed in the familiarization and will be generated (15-18 times) after the end of the voluntary contractions protocol of the subsequent sessions. An electrical stimulator device will be used. Parameters will be verified using a digital oscilloscope. The device will be connected to cables that will be connected to two pairs of 25 cm2 adhesive electrodes. The first distal electrode will be placed at 80% of the line between the anterior superior iliac spine (ASIS) and the space where the medial ligament is located. The proximal electrode will be placed in the corresponding motor point, identified with a pen type electrode, in the vastus medialis. The other distal electrode will be positioned 2/3 of the line that forms from the ASIS to the lateral side of the patella, while the proximal electrode will be placed at the motor point, identified with a pen type electrode, in the muscular belly of the vastus lateralis. It will be used a pulsed current: frequency = 100 Hz, pulse duration = 400 μs, rise time = 3 s, ON time = 4 s, decay time = 3 s, and off time = 1 min. The intensity used will be the one obtained in the familiarization, or greater if tolerated.
* Surface electrical activity and activation level: Surface electromyography (EMG) activity of vastus lateralis, vastus medialis, and rectus femoris will be recorded bipolarly by two rounded electrodes of silver chloride, each measuring 20 mm in diameter and having a recording diameter of 10 mm and separated by an inter-electrode distance (center to center) of 20 mm. The electrodes will be positioned longitudinally in the muscle belly, and a reference electrode will be attached to the patella of the contralateral lower limb. As in the case of NMES electrodes, a marking will be made to ensure that in the following sessions the electrodes will be placed accordingly. The impedance reduction (<5 kΩ) between the two electrodes will be obtained by abrasion of the skin with emery paper and cleaning with alcohol. EMG signals will be amplified with a bandwidth frequency of 15 Hz to 5.0 kilohertz (common mode rejection rate = 90 decibels, impedance = 100 milliohms, gain = 1000).
* Muscle architecture: Muscle thickness, pennation angle and fascicular length will be obtained in rest and during MVIC and NMES using a portable ultrasound in B mode with a linear transducer of 7.5 megahertz . Depth, gain, compression and ultrasound settings will be kept constant between assessments and from one patient to another. For each muscle, three videos will be obtained and the mean values will be used for statistical analysis. For better reproducibility, the evaluator will remove and reposition the transducer at the marked location. The videos will be stored on the device and then transferred to a computer for processing in specific softwares. The videos will be obtained with the transducer positioned in the longitudinal plane of the muscle, keeping it in parallel with the direction of the fascicles. Proper alignment of the transducer will be achieved when multiple fascicles are showed without interruption. Rectus femoris, vastus intermedius, vastus lateralis, vastus medialis will be evaluated, respectively, in the percentages 50%, 60% and 75% (proximal to distal) of the distance between the medial aspect of the anterior superior iliac spine and the superior border of the patella, as adapted from Blazevich et al. (2006). The rectus femoris and the vastus intermedius will be visualized on the anterior aspect of the thigh, the vastus lateralis will be visualized by moving the transducer 5 cm in the lateral direction from the midline and the vastus medialis will be visualized with the transducer 3 cm onto the medial direction of the thigh. The pennation angle is the angle formed between the echo of the deep aponeurosis of the muscles and the echo of the space between the fascicles, as measured 3 to 4 mm above the deep aponeurosis of the muscles. The fascicular length will be considered as the total length of the muscle fiber, however, because the fascicles are too long to be measured from the origin to the insertion, the estimated length will be obtained from the formula of Blazevich et al. (2006), which uses as variables the muscle thickness, the angle of the fascicle and the angle between the superficial and deep aponeurosis.
* Tendon-aponeurosis complex elongation: The myotendinous elongation will be estimated by the displacement of the deep aponeurosis. For the calculation will be used the recordings acquired for analysis of the muscular architecture. However, unlike the static nature of the data of the previous topic, this variable uses a dynamic approach, since the point (P) will be used as the contact point (insertion) of a fascicle in the deep aponeurosis at rest and the displacement of P when considering its final position during a maximum contraction. Therefore, the displacement of P (dL) is considered an indication of the elongation of the deep aponeurosis and the distal tendon.
* Tendon properties: The resting length of the patellar tendon will be measured by tracing its path with the ultrasound transducer in the longitudinal (sagittal) plane, starting from the patellar insertion to the insertion at the tibia, along the posterior surface of the tendon. The central region of the transducer will be placed in each of the tendon insertions (considering its posterior surface) and then a mark on the skin will be made at that point and a measuring tape will be used for the tendon length measurement. The cross-sectional area of the patellar tendon will be calculated from axial plane images at 25%, 50% and 75% of its length (at rest). The calculation of tendon force will use the ratio of the estimated total knee extension moment (corrected for the activation of the biceps femoris muscle obtained by electromyography) by the internal moment arm, which will be estimated by individually measuring the length of the femur, according to the equation of Visser et al (1990). Tendon stress will be calculated by the force ratio applied to the tendon by its cross-sectional area. The strain in the tendon will be calculated using the change in length over the original length (ΔL / Lo) and will be expressed as a percentage. The Young's modulus, or elastic modulus, will be obtained by dividing the stress by the strain. The tendinous stiffness will be calculated by dividing the force applied to the tendon by the elongation generated in its length. As the length of the transducer does not allow the entire visualization of the patellar tendon, a hypoallergenic echo-absorbent adhesive tape will be placed in the center of the tendon for reference. Thus, images will be obtained from the tape to the proximal insertion and then departing from the tape to the distal insertion. Images will be reconstructed for measurement. The deformation will be defined as the change in the length between the patella and the tibia, which will be measured frame-by-frame.

ELIGIBILITY:
Inclusion Criteria:

* Legal adult up to 35
* Males
* Body Massa Index: ≥ 18,5 - 24,9 kg/m²)
* International Physical Activity Questionnaire: active (but not engaged in systematic strengthening training of lower limbs)

Exclusion Criteria:

* Pain, edema, dermic injury, deformity or amputation in the body parts to be examined;
* Conditions that may affect the studied variables, such as ankylosing spondylitis, rheumatoid arthritis, diabetes mellitus, familial hypercholesterolemia, another neuromuscular disease, congestive heart failure, chronic obstructive pulmonary disease, and chronic alcoholism.
* Conditions that may affect cooperation, such as cognitive or psychiatric disease and chemical dependence.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Dynamometry: Isometric evoked torque | The peak torque of a seven-second contraction assessed in four different lower limb positions.
  Torque generated in a dynamometer during neuromuscular electrical stimulation of the quadriceps femoris muscle.
Dynamometry: Maximal Voluntary Isometric Contraction | The peak torque of a seven-second contraction assessed in four different lower limb positions.
  Torque generated in a dynamometer during maximal voluntary isometric contraction of the quadriceps femoris muscle.
Ultrasonography: Muscle Thickness | Change from rest to the end of a seven-second ramp contraction.
  Thickness of each component of the quadriceps muscle assessed by ultrasonography both in rest and during voluntary and evoked contraction.
Ultrasonography: Pennation angle | Change from rest to the end of a seven-second ramp contraction.
  Ultrasonography will be used to assess the Angle formed by the fascicles and the deep aponeurosis in which they insert both in rest and during voluntary and evoked contraction.
Ultrasonography: Fascicle length | Change from rest to the end of a seven-second ramp contraction.
  Ultrasonography will be used to assess the fascicle length both in rest and during voluntary and evoked contraction.
Ultrasonography: Tendon-aponeurosis complex elongation | Change from rest to the end of a seven-second ramp contraction.
  Ultrasonography will be used to assess the tendon-aponeurosis complex elongation of each component of the quadriceps muscle from rest to maximal voluntary and evoked contraction.
Ultrasonography: Patellar tendon properties | Change from rest to the end of a seven-second ramp contraction.
  Variables assessed from the elongation of the patellar tendon during maximal voluntary and evoked contraction.
Surface electromyography | Change from rest to the end of a seven-second ramp contraction.
  Electromyographic activity of each superficial component of the quadriceps muscle both in rest and during voluntary.

SECONDARY OUTCOMES:
Maximal tolerated intensity | The mean of the 12 repetitions in each session (1 per week, total of 4 sessions).
  Intensity or amplitude (in milliamps) of the electrical pulse during neuromuscular electrical stimulation.
Muscle fatigue | The mean of 3 repetitions in the beginning and in the end of each session (1 per week, total of 4 sessions).
  Changes in neuromuscular activation at the beginning and at the end of each session.

CONTACTS AND LOCATIONS:
Overall Officials: João LQ Durigan, PhD, Study Director — University of Brasilia
Locations (1):
- University of Brasília, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bax L, Staes F, Verhagen A. Does neuromuscular electrical stimulation strengthen the quadriceps femoris? A systematic review of randomised controlled trials. Sports Med. 2005;35(3):191-212. doi: 10.2165/00007256-200535030-00002. PMID 15730336
- [Background] Blazevich AJ, Gill ND, Zhou S. Intra- and intermuscular variation in human quadriceps femoris architecture assessed in vivo. J Anat. 2006 Sep;209(3):289-310. doi: 10.1111/j.1469-7580.2006.00619.x. PMID 16928199
- [Background] Canepari M, Pellegrino MA, D'Antona G, Bottinelli R. Skeletal muscle fibre diversity and the underlying mechanisms. Acta Physiol (Oxf). 2010 Aug;199(4):465-76. doi: 10.1111/j.1748-1716.2010.02118.x. Epub 2010 Mar 24. PMID 20345415
- [Background] de Ruiter CJ, Hoddenbach JG, Huurnink A, de Haan A. Relative torque contribution of vastus medialis muscle at different knee angles. Acta Physiol (Oxf). 2008 Nov;194(3):223-37. doi: 10.1111/j.1748-1716.2008.01888.x. Epub 2008 Aug 9. PMID 18691348
- [Background] Deley G, Babault N. Could Low-Frequency Electromyostimulation Training be an Effective Alternative to Endurance Training? An Overview in One Adult. J Sports Sci Med. 2014 May 1;13(2):444-50. eCollection 2014 May. PMID 24790503
- [Background] Doucet BM, Lam A, Griffin L. Neuromuscular electrical stimulation for skeletal muscle function. Yale J Biol Med. 2012 Jun;85(2):201-15. Epub 2012 Jun 25. PMID 22737049
- [Background] Dudley-Javoroski S, McMullen T, Borgwardt MR, Peranich LM, Shields RK. Reliability and responsiveness of musculoskeletal ultrasound in subjects with and without spinal cord injury. Ultrasound Med Biol. 2010 Oct;36(10):1594-607. doi: 10.1016/j.ultrasmedbio.2010.07.019. PMID 20800961
- [Background] Duffell LD, Dharni H, Strutton PH, McGregor AH. Electromyographic activity of the quadriceps components during the final degrees of knee extension. J Back Musculoskelet Rehabil. 2011;24(4):215-23. doi: 10.3233/BMR-2011-0298. PMID 22142710
- [Background] Fahey TD, Harvey M, Schroeder RV, Ferguson F. Influence of sex differences and knee joint position on electrical stimulation-modulated strength increases. Med Sci Sports Exerc. 1985 Feb;17(1):144-7. PMID 3872399
- [Background] Gondin J, Guette M, Ballay Y, Martin A. Electromyostimulation training effects on neural drive and muscle architecture. Med Sci Sports Exerc. 2005 Aug;37(8):1291-9. doi: 10.1249/01.mss.0000175090.49048.41. PMID 16118574
- [Background] Kawakami Y, Abe T, Fukunaga T. Muscle-fiber pennation angles are greater in hypertrophied than in normal muscles. J Appl Physiol (1985). 1993 Jun;74(6):2740-4. doi: 10.1152/jappl.1993.74.6.2740. PMID 8365975
- [Background] Arts IM, Pillen S, Schelhaas HJ, Overeem S, Zwarts MJ. Normal values for quantitative muscle ultrasonography in adults. Muscle Nerve. 2010 Jan;41(1):32-41. doi: 10.1002/mus.21458. PMID 19722256
- [Background] Pette D, Vrbova G. The Contribution of Neuromuscular Stimulation in Elucidating Muscle Plasticity Revisited. Eur J Transl Myol. 2017 Feb 24;27(1):6368. doi: 10.4081/ejtm.2017.6368. eCollection 2017 Feb 24. PMID 28458806
- [Background] Poulsen JB, Moller K, Jensen CV, Weisdorf S, Kehlet H, Perner A. Effect of transcutaneous electrical muscle stimulation on muscle volume in patients with septic shock. Crit Care Med. 2011 Mar;39(3):456-61. doi: 10.1097/CCM.0b013e318205c7bc. PMID 21150583
- [Background] Visscher RMS, Rossi D, Friesenbichler B, Dohm-Acker M, Rosenheck T, Maffiuletti NA. Vastus medialis and lateralis activity during voluntary and stimulated contractions. Muscle Nerve. 2017 Nov;56(5):968-974. doi: 10.1002/mus.25542. Epub 2017 Mar 23. PMID 28029696
- [Background] Vivodtzev I, Pepin JL, Vottero G, Mayer V, Porsin B, Levy P, Wuyam B. Improvement in quadriceps strength and dyspnea in daily tasks after 1 month of electrical stimulation in severely deconditioned and malnourished COPD. Chest. 2006 Jun;129(6):1540-8. doi: 10.1378/chest.129.6.1540. PMID 16778272
- [Derived] Cavalcante JGT, Marqueti RC, Geremia JM, de Sousa Neto IV, Baroni BM, Silbernagel KG, Bottaro M, Babault N, Durigan JLQ. The Effect of Quadriceps Muscle Length on Maximum Neuromuscular Electrical Stimulation Evoked Contraction, Muscle Architecture, and Tendon-Aponeurosis Stiffness. Front Physiol. 2021 Mar 29;12:633589. doi: 10.3389/fphys.2021.633589. eCollection 2021. PMID 33854439